CLINICAL TRIAL: NCT03163953
Title: Survey and Promoting Physical Activity in Employees and Entrepreneurial Projects of Software Park Thailand Under the Office of Science and Technology (NSTDA.)
Brief Title: Promoting Physical Activity and Break in Office Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chutima Jalayondeja, Principal investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MU-CIRB 2016/052.0804
Record Dates: First submitted 2017-05-11; First posted 2017-05-23 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: Physical Activity; Sedentary Lifestyle; Office Workers
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Tissue Polypeptide Antigen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not involve with the process of subject recruitment and allocation into three groups throughout the 6 months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TPAG with long break (Experimental): PA coaching based on TPAG and long break or break 15 minutes for every 2 hours (TPAG with LB)
  Interventions: Behavioral: TPAG with long break
- TPAG with short break (Experimental): PA coaching based on TPAG and short break or break 1-2 minutes for every 1 hours (TPAG with SB)
  Interventions: Behavioral: TPAG with short break
- Control (Other): No intervention
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: TPAG with long break — PA coaching based on Thai Physical Activity Guideline (TPAG) and long break or break 15 minutes for every 2 hours (TPAG with LB)
  Arms: TPAG with long break
Behavioral: TPAG with short break — PA coaching based on TPAG and short break or break 1-2 minutes for every 1 hours (TPAG with SB)
  Arms: TPAG with short break
Other: Control — No intervention
  Arms: Control

SUMMARY:
This study will determine the effect of physical activity promotion based on Thai Physical Activity Guideline (TPAG) and break in workplace sitting on physical activity level, physical fitness, body compositions, cognitive functions and cardiometabolic biomarkers in office workers at Software Park Thailand under the Office of Science and Technology (NSTDA). There are two intervention including physical activity (PA) coaching based on TPAG and break in workplace sitting. The investigators will coach participants for promoting daily active life and participating to monthly exercise programs. The participants will be assign to break in sitting during daily work.

DETAILED DESCRIPTION:
Objective: this study will determine the effect of physical activity promotion based on Thai Physical Activity Guideline (TPAG) and break in workplace sitting on physical activity level, physical fitness, body compositions, cognitive functions and cardiometabolic biomarkers in office workers at Software Park Thailand under the Office of Science and Technology (NSTDA).

Study design: an experimental study Interventions: there are two intervention including physical activity (PA) coaching based on TPAG and break in workplace sitting. We coach them for promoting daily active life and participating to monthly exercise programs. They will assign to break in sitting during daily work.

Methods: The office workers at Software Park Thailand under the Office of Science and Technology (NSTDA) will be invited to participate in this study. The participants are a convenience sample. The inclusion criteria are: a) age 20-60 years, b) body mass index (BMI) ≤23, c) sitting for work more than 8 hours/day, and d) physical inactivity according to the PA recommendation of the World Health Organization (WHO). The participants will be divided into three groups as the following.

Experiment 1: 30 subjects will receive PA coaching based on TPAG and long break or break 15 minutes for every 2 hours (TPAG with LB) Experiment 2: 30 subjects will receive PA coaching based on TPAG and short break or break 1-2 minutes for every 1 hours (TPAG with SB) Control group: 30 subjects will not receive interventions (control). Demographics are measured by the online self-reported questionnaire. The participants will be assessed physical activity level, physical fitness, body compositions, cognitive function and cardiometabolic biomarkers at baseline, 2-and 6-month after intervention. PA level is measured by the questionnaires and the 6-step ladder of TPAG for PA promotion. Physical fitness includes muscles strength and endurance, range of motion (ROM) and the 3-minute step test measured by the non invasive hemodynamic monitors. Body compositions comprise of BMI, waist circumference, waist to height ratio and body fat measured by the Bioelectrical Impedance Analysis. Cognitions comprise of stroop color and word test, verbal fluency, digit span test and simple reaction time test. The blood test is used to detect the cardiometabolic biomarkers such as fasting blood glucose, glycated hemoglobin (HbA1c), HDL, LDL and total cholesterol.

Statistical analysis: The statistical package for social sciences (SPSS) version 21.0 will be used for data analysis. Two-way mixed model will be used for determining the effect of PA promotion based on TPAG and break in workplace sitting on health outcomes among office workers.

ELIGIBILITY:
Inclusion Criteria:

* Works related to computer or office workers who works more than 2 years
* BMI more than 23
* Have a sedentary lifestyle or insufficient physical activity (level 0-1 evaluate by 6-stairs of Thailand Physical Activity Guideline)
* Thai people who have a good communication skill in the Thai language

Exclusion Criteria:

* Have a communication or cognition problem evaluate by Thai Mental Stat Examination
* Have a body disability
* Doctor advice don't exercise or have a fail result from Physical Activity Readiness Questionnaire
* Have a pain evaluate by Numeric Rating Scale more than 5

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-05 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Change fasting blood glucose | Change from baseline blood glucose at 6 months
  Blood sample test to measure fasting blood glucose (mg/dL)

SECONDARY OUTCOMES:
Change physical activity | Change from baseline physical activity at 6 months
  Questionnaire to measure physical activity (kcal/week)
Change cholesterol | Change from baseline HDL cholesterol at 6 months
  Blood sample test to measure HDL cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Chutima Jalayondeja, Dr.P.H., Principal Investigator — Faculty of Physical Therapy, Mahidol University, Thailand
Locations (1):
- Mahidol University, Salaya, Nakon Prothom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available for other researchers after the end of the study.

REFERENCES:
- [Result] Jalayondeja C, Jalayondeja W, Vachalathiti R, Bovonsunthonchai S, Sakulsriprasert P, Kaewkhuntee W, Bunprajun T, Upiriyasakul R. Cross-Cultural Adaptation of the Compendium of Physical Activity: Thai Translation and Content Validity. J Med Assoc Thai. 2015 Jun;98 Suppl 5:S53-9. PMID 26387412
- [Result] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120
- [Result] Jalayondeja C, Jalayondeja W, Mekhora K, Bhuanantanondh P, Dusadi-Isariyavong A, Upiriyasakul R. Break in Sedentary Behavior Reduces the Risk of Noncommunicable Diseases and Cardiometabolic Risk Factors among Workers in a Petroleum Company. Int J Environ Res Public Health. 2017 May 9;14(5):501. doi: 10.3390/ijerph14050501. PMID 28486414